CLINICAL TRIAL: NCT00004449
Title: Randomized Study of Intensive One-on-one Behavioral Treatment Versus Individualized Parent Training in Preschool Aged Children With Autism
Brief Title: Randomized Study of Intensive One-on-one Behavioral Treatment for Preschool Aged Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tristram Smith, Ph.D., Professor of Pediatrics, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01MH048863 (NIH); R01MH048863 (NIH); UCLA-HSPC-G930506611
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Autistic Disorder
Keywords: autism; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Autistic Disorder; Neurologic Manifestations; Mental Disorders; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: intensive one-on-one behavioral treatment — Up to 40 hours per week of one-to-one intervention based on applied behavior analysis
Behavioral: Individualized in home parent training — Offered to subjects at some sites, involved 3+ months of individualized training for parents on applied behavior analysis intervention

SUMMARY:
OBJECTIVES: I. Determine the effectiveness of intensive one-on-one behavioral treatment in the home or neighborhood compared with at home, individualized, parent training in preschool aged children with autism.

II. Identify intake measures that predict differences in outcome between subjects in the experimental group.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. Children are randomized to receive either 35 hours of intensive one-on-one behavioral treatment in the home and neighborhood for 2 years or individualized, in home parent training for 6 months.

A common group of tests to evaluate autism are administered at intake, 12 and 24 months into treatment, and when patients reach age 6.

ELIGIBILITY:
INCLUSION CRITERIA:

--Disease Characteristics--

Diagnosis of autism based on the Autism Diagnostic Interview using the ICD-10 research criteria

Ratio IQ score greater than 35 determined from the Bayley Scales of Infant Development

--Patient Characteristics--

Other:

Must reside within 60 km (37.5 miles) of a treatment site

EXCLUSION CRITERIA:

Severe medically induced limitations defined as:

* Any condition requiring prosthetic devices (e.g., blindness, deafness, or cerebral palsy)
* Any illness that has prevented or would prevent a subject from participating in 30 hours a week of treatment for six consecutive weeks or more (e.g., metastasized cancer or end stage renal disease)
* Any known genetic disorder (e.g., Fragile X, PKU, or Down Syndrome)
* Any other disorder that rules out autism according to ICD-10 criteria (e.g., Rett's Syndrome)

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 1998-05; Primary Completion 2004-09 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Wechsler Preschool and Primary Scales of Intelligence, 3rd ed. | yearly for up to 4 years
  IQ
Bayley Scales of Infant Development | yearly for up to 4 years
  Alternate cognitive test administered to participants who did not achieve basal on WPPSI-III

SECONDARY OUTCOMES:
Merrill-Palmer Scale of Mental Tests | yearly for up to 4 years
  Nonverbal cognitive skills
Reynell Developmental Language Scales | yearly for up to 4 years
  Language comprehension and expressive language
Vineland Adaptive Behavior Scales - Survey Edition | yearly for up to 4 years
  Parent interview on child's adaptive functioning

CONTACTS AND LOCATIONS:
Overall Officials: Tristram Smith, Ph.D., Study Director — University of Rochester

REFERENCES:
- [Result] Cohen H, Amerine-Dickens M, Smith T. Early intensive behavioral treatment: replication of the UCLA model in a community setting. J Dev Behav Pediatr. 2006 Apr;27(2 Suppl):S145-55. doi: 10.1097/00004703-200604002-00013. PMID 16685181
- [Result] Sallows GO, Graupner TD. Intensive behavioral treatment for children with autism: four-year outcome and predictors. Am J Ment Retard. 2005 Nov;110(6):417-38. doi: 10.1352/0895-8017(2005)110[417:IBTFCW]2.0.CO;2. PMID 16212446
- [Result] Hayward D, Eikeseth S, Gale C, Morgan S. Assessing progress during treatment for young children with autism receiving intensive behavioural interventions. Autism. 2009 Nov;13(6):613-33. doi: 10.1177/1362361309340029. PMID 19933766